CLINICAL TRIAL: NCT05667415
Title: Clinical Study of Disulfiram Combined With Cisplatin in the Treatment of Advanced Gastric Cancer
Brief Title: Treatment of Advance Gastric Cancer With Disulfiram
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: College of Pharmaceutical Sciences at Zhejiang University (Unknown); The Innovation Institute for Artificial Intelligence in Medicine, Zhejiang University (Unknown)
Responsible Party: Principal Investigator, Zhang Xiaofeng,MD, chief physician, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221212
Record Dates: First submitted 2022-12-12; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Chemotherapy；Advanced Gastric Cancer；Cisplatin；Disulfiram
MeSH Terms: interventions — Disulfiram; Cisplatin

STUDY DESIGN:
Intervention Model Description: Combination regimen of disulfiram and cisplatin for gastric cancer and standard cisplatin regimen for gastric cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- disulfiram and cisplatin (Experimental): Cisplatin combined with disulfiram chemotherapy
  Interventions: Drug: disulfiram and cisplatin
- standard cisplatin (Active Comparator): Cisplatin chemotherapy alone
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: disulfiram and cisplatin — on the first day of treatment, patients were given intravenous drip of 80mg/m2 cisplatin, and 21 days was a course of treatment, lasting for 6 courses. Take 400mg disulfiram orally every day, and continue to use it until the end of chemotherapy. According to the patient's tolerance to disulfiram, the dose of disulfiram can be re-evaluated during the treatment, and the lowest dose is 125mg per day. The clinical symptoms, signs and adverse reactions of patients were observed, and the treatment effect of patients was evaluated after two consecutive cycles with 3 weeks as a cycle.
  Arms: disulfiram and cisplatin
Drug: cisplatin — on the first day of treatment, patients were given 80mg/m2 cisplatin intravenously, and 21 days was a course of treatment, lasting for 6 courses.
  Arms: standard cisplatin

SUMMARY:
Chemotherapy is generally needed for advanced gastric cancer, and cisplatin is the main chemotherapy drug. However, there are many adverse reactions, including bone marrow suppression, gastrointestinal reactions, renal toxicity and neurotoxicity. These adverse reactions can affect the comfort and compliance of patients during treatment. At present, it is necessary to reduce adverse reactions of cisplatin and increase the chemotherapy sensitivity of gastric cancer to cisplatin. Recent studies have found that disulfiram has a potential anti-tumor effect. The disulfiram has shown significant in vivo and in vitro anti-tumor activity in preclinical studies, and has become a potential candidate drug for tumor treatment as an adjuvant in various clinical trials. In this clinical study, cisplatin combined with disulfiram is mainly used to treat advanced gastric cancer.

DETAILED DESCRIPTION:
Chemotherapy is generally needed for advanced gastric cancer, and cisplatin is the main chemotherapy drug. However, there are many adverse reactions, including bone marrow suppression, gastrointestinal reactions, renal toxicity and neurotoxicity. These adverse reactions can affect the comfort and compliance of patients during treatment. At present, it is necessary to reduce adverse reactions of cisplatin and increase the chemotherapy sensitivity of gastric cancer to cisplatin. Recent studies have found that disulfiram has a potential anti-tumor effect. The disulfiram has shown significant in vivo and in vitro anti-tumor activity in preclinical studies, and has become a potential candidate drug for tumor treatment as an adjuvant in various clinical trials. In this clinical study, cisplatin combined with disulfiram is mainly used to treat advanced gastric cancer.Subjects were randomized in a 1:1 ratio, one group being the control group and the other group being the observation group. Control group: On the first day of treatment, the patients were given intravenous drip of 80mg/m2 cisplatin, 21 days as a course of treatment, lasting for six courses. Observation group: On the first day of treatment, the patients were given intravenous drip of 80mg/m2 cisplatin, 21 days as a course of treatment, lasting for six courses. Disulfiram 400mg was given orally daily and continued until the end of the chemotherapy course. Based on the patient's tolerance to disulfiram, the disulfiram dose may be reassessed during treatment with a minimum oral dose of 125mg per day. The clinical symptoms, signs and adverse reactions were observed in the patients, and the treatment effect was evaluated after three weeks as a cycle and two cycles.

ELIGIBILITY:
1. Inclusion criteria: ① Age ≥18 years old; ② Gastric cancer is confirmed through gastroscopy biopsy; ③ The patient meets the relevant diagnostic criteria in People's Republic of China (PRC) Health Industry Standards: Diagnostic Criteria for Gastric Cancer, and has reached the level of stage III and IV futures, and the patient refuses to receive surgical treatment; ④ Estimated survival time > 3 months; ⑤ Without any chemotherapy treatment or more than one month from the end of the last chemotherapy course; ⑥Karnofsky functional status score ≥ 60;
2. Exclusion criteria: ① patients who had allergic reaction to therapeutic drugs; ② patients with other types of cancer; ③ Patients with severe diseases of heart, liver, kidney, etc.; (4) gastrointestinal dysfunction or unable to oral medication.
3. Shedding/eliminating criteria: exiting in the midway; Lost to follow-up during the follow-up period; Treatment was not continued according to the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | every 6 weeks
  The tumor lesion in our patient completely resolved and lasted for ≥4 weeks, and no new lesion appeared
Partial response (PR) | every 6 weeks
  the overall reduction in the longest diameter of the tumor focus is > 50% and it can be maintained for at least 4 weeks, with no new focus emerging
Stable disease (SD) | every 6 weeks
  the overall reduction or increase of the longest diameter of the tumor lesion is < 50% or < 25%, and the duration is > 4 weeks; no new lesion appears
Disease progression (PD) | every 6 weeks
  the combined increase in the longest diameter of the tumor lesion is ≥25%, or a new lesion appears

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No